CLINICAL TRIAL: NCT00800735
Title: An Open-label, Multicenter Protocol Providing Pegylated-interferon Alfa-2a (PEGASYS®) as Monotherapy or in Combination With Ribavirin (COPEGUS®) for Patients With Chronic Hepatitis C Who Have Participated in Previous Roche or Roche Partner Protocols
Brief Title: A Study of PEGASYS (Pegylated-interferon Alfa-2a) With or Without Ribavirin in Patients With Chronic Hepatitis C Who Have Participated in Previous Roche or Roche Partner Protocols
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV21928; 2008-002022-10
Record Dates: First submitted 2008-10-23; First posted 2008-12-02 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (1):
- Pegylated-interferon alfa-2a plus ribavirin (Experimental): Participants received pegylated-interferon alfa-2a 180 µg/week subcutaneously plus ribavirin 1000 mg/day orally for patients weighing < 75 kg or 1200 mg/day for patients weighing ≥ 75 kg for 48 weeks.
  Interventions: Drug: Pegylated-interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated-interferon alfa-2a — Pegylated-interferon alfa-2a was administered subcutaneously once weekly.
  Other Names: PEG-IFN alfa-2a; Pegasys
Drug: Ribavirin — Participants received ribavirin with food, as the bioavailability of ribavirin is increased when taken with food. Ribavirin was administered as split doses, that is, 2 doses were given 12 hours apart, 1 in the morning and 1 in the evening. Participants received either 1000 or 1200 mg ribavirin per day according to body weight: 400 mg (2 tablets) in the morning and 600 mg (3 tablets) in the evening for participants weighing < 75 kg or 600 mg (3 tablets) in the morning and 600 mg (3 tablets) in the evening for participants weighing ≥ 75 kg.
  Other Names: Copegus; Ro 20-9963

SUMMARY:
This single arm study will provide treatment or re-treatment with PEGASYS as monotherapy or in combination with ribavirin (Copegus), to patients with chronic hepatitis C (CHC) who have participated in a previous Roche or Roche partner protocol where access to treatment or re-treatment was promised or deemed appropriate following completion of the original protocol ('donor' protocol). Patients who qualify for treatment or re-treatment will begin PEGASYS monotherapy, at a maximum dose of 180 µg weekly, or combination therapy with Copegus, 800-1200 mg daily, as continuation of treatment after the wash-out period defined in their donor protocol. PEGASYS treatment is not to exceed the approved treatment duration of 48 weeks in genotype G1 with a treatment-free follow up period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Chronic hepatitis C (CHC) patients with compensated liver disease (Child-Pugh A) who have participated in a donor protocol where access to treatment or re-treatment with PEGASYS monotherapy or in combination with Copegus was promised or deemed appropriate after completion of the donor protocol.

Exclusion Criteria:

* Evidence of decompensated liver disease (Child B or C cirrhosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (11):
  - Sacramento, California
  - San Francisco, California
  - Lutherville, Maryland
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Providence, Rhode Island
  - Nashville, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah
- Vienna, Austria
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- Clichy, France
- Germany (3):
  - Berlin
  - Cologne
  - Frankfurt am Main
- Spain (4):
  - Badalona
  - Barcelona
  - Madrid
  - Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegylated-interferon Alfa-2a Plus Ribavirin
Started | 30
Completed | 16
Not Completed | 14
Not completed — Administrative/Other | 2
Not completed — Insufficient Therapeutic Response | 2
Not completed — Violation of Selection Criteria at Entry | 7
Not completed — Withdrew Consent | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated-interferon Alfa-2a Plus Ribavirin
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2
  Caucasian | 28
Height [Mean (Standard Deviation); unit: cm] | 170.0 (7.28)
Weight [Mean (Standard Deviation); unit: kg] | 76.97 (16.146)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.53)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event.
Description: An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline through 24 weeks after the end of treatment (up to 72 weeks)
Population: All enrolled patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Pegylated-interferon Alfa-2a Plus Ribavirin
Number analyzed (Participants) | 30
Percentage of participants | 80.0

ADVERSE EVENTS:
Time Frame: Adverse events from the beginning of treatment up to 24 weeks after the end of treatment were reported.
Description: Safety population: All enrolled participants.
Arm/Group | Pegylated-interferon Alfa-2a Plus Ribavirin
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated-interferon Alfa-2a Plus Ribavirin (N=30)
Retinal haemorrhage (Eye disorders) | 1
Conjunctivitis viral (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Prothrombin time prolonged (Investigations) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated-interferon Alfa-2a Plus Ribavirin (N=30)
Anaemia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 4
Hyperthyroidism (Endocrine disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 5
Chills (General disorders) | 7
Fatigue (General disorders) | 16
Influenza like illness (General disorders) | 5
Pyrexia (General disorders) | 4
Bronchitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.